CLINICAL TRIAL: NCT06099067
Title: Harmonizing RCT-Duplicate Emulations: A Real World Replication Program Analyzing Three Clinical Trials, CANVAS, LEADER, and SAVOR TIMI in Type 2 Diabetes Mellitus
Brief Title: Harmonizing RCT-Duplicate Emulations In A Real World Replication Program (HARRP)
Acronym: HARRP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00345
Record Dates: First submitted 2023-04-06; First posted 2023-10-25 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Clinical Trial; Emulation; Epidemiology; Type 2 Diabetes; Regulatory; Real World Evidence; Real World Data
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Dipeptidyl-Peptidase IV Inhibitors; Liraglutide; saxagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CANVAS Canagliflozin: CANVAS expousre Group
  Interventions: Drug: Canagliflozin
- CANVAS DPP4i: CANVAS reference Group
  Interventions: Drug: DPP4 inhibitor
- LEADER Liraglutide: LEADER exposure Group
  Interventions: Drug: Liraglutide
- LEADER DPP4i: LEADER reference Group
  Interventions: Drug: DPP4 inhibitor
- SAVOR-TIMI Saxagliptin: SAVOR-TIMI exposure Group
  Interventions: Drug: Saxagliptin
- SAVOR-TIMI 2nd generation Sulfonylurea: SAVOR-TIMI reference Group
  Interventions: Drug: 2nd generation Sulfonylurea

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin dispensing claim is used as the exposure drug in CANVAS replication
  Groups: CANVAS Canagliflozin
Drug: DPP4 inhibitor — DPP4 inhibitor dispensing claim is used as the reference drug in CANVAS and LEADER replications
  Groups: CANVAS DPP4i; LEADER DPP4i
Drug: Liraglutide — Liraglutide dispensing claim is used as the Exposure drug in LEADER replication
  Groups: LEADER Liraglutide
Drug: Saxagliptin — Saxagliptin dispensing claim is used as the Exposure drug in SAVOR-TIMI replication
  Groups: SAVOR-TIMI Saxagliptin
Drug: 2nd generation Sulfonylurea — 2nd generation Sulfonylurea dispensing claim is used as the Exposure drug in SAVOR-TIMI replication
  Groups: SAVOR-TIMI 2nd generation Sulfonylurea

SUMMARY:
Replication of three clinical trial emulations CANVAS, LEADER, and SAVOR TIMI that form part of the RCT-Duplicate initiative, sponsored by the FDA and delivered by the Brigham and Women's Hospital and Harvard Medical School. AstraZeneca will use the Instant Health Data platform PANALGOS (IHD) for the analyses.

DETAILED DESCRIPTION:
RCT-duplicate (RCT-D) is an initiative led by the Brigham and Women's Hospital and Harvard Medical School, that selected 30 clinical trials as part of an empirical experiment where these trials would be emulated using RWD. AstraZeneca will replicate three emulations CANVAS, LEADER, and SAVOR TIMI from among the 30 plus clinical trials analyzed in RCT-D. These clinical trials assess type 2 diabetes mellitus drugs. The replications will be conducted on the Instant Health Data PANALGOS (IHD) platform to assess these studies in two claims databases Optum and IBM Watson Market Scan. The aim is to recreate these three emulations to investigate the reproducibility of the emulations, increase transparency and better understand the process of trial emulations; and where possible, contribute with potential improvements to the RCT-D framework.

ELIGIBILITY:
The Eligibility Criteria for CANVAS, LEADER and SAVOR-TIMI are replicated

Please see the Criteria for each under:

* CANVAS: https://clinicaltrials.gov/ct2/show/NCT03936010
* LEADER: https://clinicaltrials.gov/ct2/show/NCT03936049
* SAVOR-TIMI: https://clinicaltrials.gov/ct2/show/NCT03936023

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus (T2DM) adult patients enrolled in the two claims databases and are eligible to be included according to the inclusion and exclusion criteria of each of the three investigated clinical trial studies: CANVAS, LEADER and SAVOR-TIMI.
  All subjects meeting the inclusion and exclusion criteria will be assessed. Remaining sample size will be dependent on the number of matched subjects in each cohort using the two data sources combined.
Sampling Method: Non-Probability Sample
Enrollment: 239990 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
3-point MACE | Follow up begins the day after drug initiation for the three investigated studies [a median of 134-167 days]
  3-point MACE: Relative hazard of composite outcome of Stroke, MI, and Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: from 05 December 2022
Access Criteria: Protocol and SAP details along with programming code to be supplied upon request via mail.

REFERENCES:
- See also: CANVAS — https://clinicaltrials.gov/ct2/show/NCT03936010
- See also: LEADER — https://clinicaltrials.gov/ct2/show/NCT03936049
- See also: SAVOR-TIMI — https://clinicaltrials.gov/ct2/show/NCT03936023
- See also: The Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00345&attachmentIdentifier=6f9731f7-7f0a-432d-bfeb-b5aaa30e1f99&fileName=Redacted_CSR_Synopsis_D1843R00345.pdf&versionIdentifier=